CLINICAL TRIAL: NCT00570284
Title: A Phase Ib Open-label, Multicenter Cross-over Study to Investigate the Effect of Food on the Rate and Extent of Oral LBH589 Absorption in Patients With Advanced Solid Tumors
Brief Title: A Study to Investigate the Effect of Food on Oral LBH589 Absorption in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2111
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-08

CONDITIONS: Cancer
Keywords: Cancer; solid tumor; food effect; HDAC inhibitor; oral; LBH589
MeSH Terms: conditions — Neoplasms | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — orally administered panobinostat at 20 mg twice weekly (core phase); orally administered panobinostat 45 mg twice weekly if 20 mg twice weekly was tolerated in Cycle 1 (extension phase)
  Other Names: Panobinostat

SUMMARY:
The primary purpose of this study is to evaluate the effect of food on oral LBH589 in adult patients with advanced solid tumors. This study will also evaluate the safety and efficacy of LBH589 in adult patients with advanced solid tumors

ELIGIBILITY:
Inclusion criteria:

* Patients with advanced solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists
* Age ≥ 18 years old
* Patients must have adequate laboratory values
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Ability to swallow capsules or tablets

Exclusion criteria:

* Patients with active central nervous system (CNS) disease or brain metastases except those who have been previously treated and have been stable for at least 3 months.
* Patients with a second primary malignancy that is currently clinically significant or requiring active intervention
* Impaired heart function or clinically significant heart disease
* Impairment of gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of LBH589
* Ongoing diarrhea
* Liver or renal disease with impaired hepatic or renal functions
* Concomitant use of any anti-cancer therapy or certain drugs
* Female patients who are pregnant or breast feeding
* Patients not willing to use an effective method of birth control

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Levels of LBH589 in the blood | every week for the first 3 weeks

SECONDARY OUTCOMES:
Efficacy, Safety and tolerability | throughout study to 28 days after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (9):
- United States (7):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Norwalk, Connecticut
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Madison, Wisconsin
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Zurich, Switzerland

REFERENCES:
- See also: Results for CLBH589B2111 on the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4924